#### NCT02013791

## Study 192371-024

Title: A Phase 2, Multi-center, Vehicle- and Sham-controlled, Randomized Study of RESTASIS® X in Patients With Moderate to Severe Dry Eye Disease

Protocol Amendment 6 Date: Jan 19, 2017

Statistical Analysis Plan (SAP) Date: June, 20, 2017

## 1. Title Page

#### STATISTICAL ANALYSIS PLAN

A Phase 2, Multicenter, Vehicle- and Sham-controlled, Randomized Study of RESTASIS® X in Patients With Moderate to Severe Dry Eye Disease

Stage 1

Protocol Number: 192371-024

Development Phase: 2

Product Name: RESTASIS® X

Study Statistician:

Sponsor: Allergan (North America)

2525 Dupont Drive Irvine, California USA

92612

+1-714-246-4500 +1-800-347-4500

This document is the property of Allergan, Inc. and may not, in full or part, be passed on, reproduced, published, distributed to any person, or submitted to any regulatory authority without the express written permission of Allergan, Inc.

# 2. Table of Contents

| 1. | Title | Page | | 1 |
|---|---|---|---|---|
| 2. | Tabl | e of Co | ntents | 2 |
| | 2.1 | List of | f Tables | 3 |
| | 2.2 | | f Figures | |
| 3. | List | | reviations and Definition of Terms | |
| 4. | | | 1 | |
| | 4.1 | | | |
| | | | Design Summary | |
| | 4.2 | _ | Objectives and Assessments | |
| | 4.3 | | lule of Activities | |
| 5. | Stati | stical M | Methodology and Study Endpoints | 18 |
| | 5.1 | Statist | tical Methods Planned in the Protocol and Determination of Sample S | Size 18 |
| | | 5.1.1 | Statistical and Analytical Plans | 18 |
| | | | 5.1.1.1 Common Conventions | 18 |
| | | | 5.1.1.2 Demographics | 20 |
| | | | 5.1.1.3 Exploratory Efficacy Analyses | 22 |
| | | | 5.1.1.4 Safety Analyses | 26 |
| | | | 5.1.1.5 Health Outcomes Data Analyses | 32 |
| | | | 5.1.1.6 Subgroup Analyses | |
| | | | 5.1.1.7 Interim Analyses | |
| | | 5.1.2 | Determination of Sample Size | |
| | 5.2 | Chang | ges in the Conduct of the Study or Planned Analyses | |
| | | 5.2.1 | Changes in the Conduct of the Study | |
| | | 5.2.2 | Changes to Analyses Prior to Database Lock | |
| 6. | Data | Handli | ing and Analysis Conventions | 34 |
| | 6.1 | Study | Treatment Conventions | 34 |
| | | 6.1.1 | Analysis Days | 34 |
| | 6.2 | Analy | vsis Visit Windows | 34 |
| | | 6.2.1 | Treatment Cycle 1 | 34 |
| | | 6.2.2 | Treatment Cycle 2 | 36 |
| | 6.3 | Missin | ng/Incomplete Date Conventions | 38 |
| | | 6.3.1 | Missing/Incomplete AE Start Date | 39 |
| | | 6.3.2 | Missing/Incomplete Medication Start Date | 39 |
| | | 6.3.3 | Missing/Incomplete AE/Medication End Date | 39 |

| 6.4 | Exploratory Efficacy Endpoint Conventions | 39 |
|---|---|---|
| | 6.4.1 Patient Symptoms (Visual Analog Scale) | 39 |
| | 6.4.2 Ocular Surface Disease Index | 40 |
| 6.5 | Safety Endpoint Conventions. | 40 |
| | 6.5.1 Adverse Events | |
| | 6.5.1.1 Missing Intensity or Relationship | |
| | 6.5.2 Clinical Laboratory Assessments | |
| | 6.5.3 Vital Signs | |
| | 6.5.5 Dilated Ophthalmic Examinations | |
| 6.6 | Health Outcomes Endpoint Conventions | |
| 6.7 | Imputed Value Listing Conventions | |
| 2.1 | List of Tables | |
| Table 3-1 | Abbreviations and Definitions of Terms | <i>6</i> |
| Гable 4-1 | Dosage/Dose Regimen – Stage 1 Dose Escalation in Patients With M<br>Severe Dry Eye Disease | oderate to |
| Гable 4-2 | Study Objectives and Corresponding Endpoints - Stage 1 | 12 |
| Гable 4-3 | Schedule of Activities - Stage 1 | 14 |
| Гable 4-4 | Schedule of Activities - Stage 2 | 16 |
| Table 5-1 | Analysis Populations – Stage 1 | 18 |
| Table 5-2 | Statistical Methodology – Stage 1 | 19 |
| Table 5-3 | Analysis Population Summaries | 20 |
| Гable 5-4 | Patient Disposition Summaries | 20 |
| Table 5-5 | Protocol Deviation Summary | 21 |
| Гable 5-6 | Demographic Summaries | 21 |
| Гable 5-7 | Medical History Summary | 21 |
| Гable 5-8 | Medication Summaries | 22 |
| Гable 5-9 | Schirmer's Tear Test Summaries. | 22 |

| Table 5-10 | Tear Film Break-Up Time Summaries | 23 |
|------------|--------------------------------------------------|----|
| Table 5-11 | Sodium Fluorescein Corneal Staining Summaries | 23 |
| Table 5-12 | Lissamine Green Conjunctival Staining Summaries | 23 |
| Table 5-13 | Patient Symptoms (Visual Analog Scale) Summaries | 24 |
| Table 5-14 | Ocular Surface Disease Index (OSDI) Summaries | 25 |
| Table 5-15 | Treatment Assessment by Investigator Summaries | 25 |
| Table 5-16 | Study Treatment Summaries | 26 |
| Table 5-17 | AE Terms | 26 |
| Table 5-18 | AE Summaries | 26 |
| Table 5-19 | Clinical Laboratory Summaries | 28 |
| Table 5-20 | Vital Signs Summaries | 28 |
| Table 5-21 | BCVA Summaries | 29 |
| Table 5-22 | Macroscopic Bulbar Hyperemia Summaries | 30 |
| Table 5-23 | Slit-lamp Biomicroscopy Summaries | 30 |
| Table 5-24 | Dilated Ophthalmic Examinations Summaries | 31 |
| Table 5-25 | Photographic Conjunctival Hyperemia Summaries | 31 |
| Table 5-26 | Intraocular Pressure Summaries | 32 |
| Table 5-27 | REFRESH PLUS Use and Compliance Summaries | 32 |
| Table 5-28 | Health Outcomes Data Summaries | 32 |
| Table 6-1 | Analysis Day Definitions | 34 |
| Table 6-2 | Analysis Visit Definitions 1 | 34 |
| Table 6-3 | Analysis Visit Definitions 2 | 34 |
| Table 6-4 | Analysis Visit Definitions 3 | 35 |
| Table 6-5 | Analysis Visit Definitions 4 | 35 |
| Table 6-6 | Analysis Visit Definitions 5 | 35 |

| Figure 4-1 | Stage 1 Study Flow – Dose Escalation In Patients With Moderate To Se Eye Disease | • |
|---|---|---|
| 2.2 | List of Figures | |
| Table 6-26 | Supplemental Dry Eye Questionnaire | 44 |
| Table 6-25 | Dilated Ophthalmic Examinations Grade | |
| | Slit-lamp Biomicroscopy Scales | |
| Table 6-23 | Vital Sign Descriptive Parameters | |
| Table 6-22 | Clinical laboratory Descriptive and Shift Table Parameters | 41 |
| Table 6-21 | Missing AE Intensity and Relationship Imputation Algorithms | 40 |
| Table 6-20 | OSDI Score Derivation | 40 |
| Table 6-19 | OSDI Questionnaire | 40 |
| Table 6-18 | Patient Symptoms (Visual Analog Scale) | 39 |
| Table 6-17 | Initial Imputed Date Algorithm | 39 |
| Table 6-16 | Imputation Scenarios | 38 |
| Table 6-15 | Analysis Visit Definitions 6 (Retreatment) | 38 |
| Table 6-14 | Analysis Visit Definitions 5 (Retreatment) | 37 |
| Table 6-13 | Analysis Visit Definitions 4 (Retreatment) | 37 |
| Table 6-12 | Analysis Visit Definitions 3 (Retreatment) | 37 |
| Table 6-11 | Analysis Visit Definitions 2 (Retreatment) | 37 |
| Table 6-10 | Analysis Visit Definitions 1 (Retreatment) | 36 |
| Table 6-9 | Analysis Visit Definitions 8 | 36 |
| Table 6-8 | Analysis Visit Definitions 7 | 36 |
| Table 6-7 | Analysis Visit Definitions 6 | 36 |

# 3. List of Abbreviations and Definition of Terms

Table 3-1 Abbreviations and Definitions of Terms

| Abbreviation/Term | Definition |
|-------------------|----------------------------------------------|
| AE | adverse event |
| BCVA | best-corrected visual acuity |
| CFB | change from baseline |
| DDE | Drug Dictionary Enhanced |
| eCRF | electronic case report form |
| F1 | |
| F2 | |
| IOP | intraocular pressure |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mITT | modified intent-to-treat |
| OSDI | Ocular Surface Disease Index |
| PK | pharmacokinetic |
| PT | preferred term |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| SOC | system organ class |
| TEAE | treatment-emergent adverse event |
| TBUT | tear film break-up time |
| VAS | visual analog scale |
| WHO | World Health Organization |

#### 4. Introduction

This statistical analysis plan (SAP) details comprehensive, technical specifications of the statistical analyses of the safety, exploratory efficacy, and health outcomes data outlined and/or specified in Protocol 192371-024 Amendment 6, dated 19 Jan 2017. Study 192371-024 is a 2-stage, Phase 2 study. A final database lock will occur after the completion of stage 2. Separate analysis plans will be prepared for the analysis of each stage. This document is the analysis plan for stage 1. Specifications of tables, figures, and data listings are contained in a separate document. The SAP for pharmacokinetic (PK) data will be prepared separately.

This document is organized into 3 main sections as follows:

- 1. Study overview
- 2. Statistical methodology and study endpoints
- 3. Data handling and analysis conventions

## 4.1 Study Design Summary

This study is a multicenter, randomized, investigator-masked, 24-week evaluation of the safety, exploratory efficacy, and pharmacokinetics of RESTASIS® X in patients with moderate to severe dry eye disease. The study is being conducted in 2 stages.

<u>Stage 1</u>: Single-dose, paired-eye comparison, dose escalation, vehicle-controlled, followed by retreatment (Cohorts 6C and 6D).

| Stage 1 will evaluate the safety and ocular and systemic pharmacokinetics of F1 |
|---|
| and F2 |









Randomization/Stratification:

Stage 1: Within each cohort, patients will be randomly assigned with respect to the eye, right or left, to receive F1 or F2 (or vehicle for Cohort 1). The contralateral eye will receive vehicle (sham for Cohort 1).



Number of Patients:

Stage 1: Stage 1 will have up to 63 patients and approximately 10 cohorts (Cohorts 1 to 6D). The anticipated numbers of patients per cohort are 3 for Cohort 1; 4 for Cohorts 2, 6C, and 6D; and 8 each for Cohorts 3 through 6B.

## 4.2 Study Objectives and Assessments

The study objective for stage 1 is presented with corresponding assessments in Table 4-2.

Table 4-2 Study Objective and Corresponding Assessments - Stage 1

| Objective Assessments | |
|---|---|
| To evaluate the safety, exploratory efficacy, and pharmacokinetics of F1 and F2 administered as a In patients with moderate to severe dry eye disease. Safety Assessments BCVA (manifest refraction at screening and exit visits) Macroscopic hyperemia assessment and slit-lamp biomi Dilated ophthalmic exam Photographic conjunctival hyperemia assessment IOP Vital signs Laboratory tests (chemistry, hematology, urinalysis) Urine pregnancy test (for females of childbearing potent) Pharmacokinetic Assessments PK assessments will be detailed in a separate PK analysis | tial) |

AE = adverse event; BCVA = best-corrected visual acuity; F1 F2 = IOP = intraocular pressure; OSDI = Ocular Surface Disease Index; PK = pharmacokinetic; TBUT = tear film break-up time; VAS = visual analog scale

## 4.3 Schedule of Activities

The schedule of activities is presented in Table 4-3 (stage 1) and Table 4-4 (stage 2). If retreatment is given at Week 12, the stage 1 retreatment schedule will be following the stage 2 retreatment schedule (see post-retreatment follow-up visits in Table 4-4).









## 5. Statistical Methodology and Study Endpoints

# 5.1 Statistical Methods Planned in the Protocol and Determination of Sample Size

This SAP for stage 1 will be approved prior to final database lock. The SAP expands the statistical section of the protocol and contains a detailed description of methods to analyze data collected in the study. The text portion of the SAP will be included in the clinical study report report as Appendix 16.1.9. Information on the PK analyses can be found in the PK data analysis plan, which is a separate document.

## 5.1.1 Statistical and Analytical Plans

#### 5.1.1.1 Common Conventions

## 5.1.1.1.1 Analysis Populations

The analysis populations will consist of patientss as defined in Table 5-1.

Table 5-1 Analysis Populations – Stage 1

| Population | Definition | Study Treatment |
|---|---|---|
| Safety | All patients who are treated | Actual received <sup>a</sup> |
| Modified intent-to- | All randomized patients who have baseline and at least 1 | D 1 1 1 1 1 1 |
| treat (mITT) | postbaseline assessment for 1 or more of the exploratory efficacy | Randomized assignment |
| | measurements | |

<sup>&</sup>lt;sup>a</sup> Patients will be summarized according to the first study treatment received or study treatment received for majority of treatment period.

## **5.1.1.1.2 Study Treatments**

The following treatment groups and cohorts are defined for stage 1 in this study:

| Cohort | Treatment Group | |
|-----------|-----------------|-----------------------------|
| Cohort 5A | RESTASIS X F1 | |
| Cohort 4 | RESTASIS X F1 | |
| Cohort 6C | RESTASIS X F1 | with retreatment at week 12 |
| Cohort 3 | RESTASIS X F1 | |
| Cohort 2 | RESTASIS X F1 | |
| Cohort 6B | RESTASIS X F2 | |
| Cohort 6D | RESTASIS X F2 | with retreatment at week 12 |
| Cohort 6A | RESTASIS X F2 | |
| Cohort 1 | Vehicle | |

Data will be analyzed by treatment group/cohort, unless otherwise specified.

## 5.1.1.1.3 Statistical Methodology

The methodologies defined in Table 5-2 apply as specified to individual endpoints defined in this SAP for stage 1.

Table 5-2 Statistical Methodology – Stage 1

| Methodology | Description |
|---|---|
| Categorical counts | Number of patients in individual categories |
| | <ul> <li>Patients with ≥ 1 qualifying event counted once per individual category</li> </ul> |
| Categorical | Number and percentage of patients in individual categories |
| descriptives | <ul> <li>○ Patients with ≥ 1 qualifying event counted once per individual category</li> </ul> |
| | <ul> <li>N1 if percentage denominator ≠ number of patients in the population (standard</li> </ul> |
| | percentage denominator) |
| | <ul> <li>N1 = patients with nonmissing value</li> </ul> |
| Continuous | N1, mean, SD, median, minimum, maximum |
| descriptives | N1 = patients with nonmissing value |
| CFB descriptives | <ul> <li>Continuous descriptives for baseline, postbaseline, and CFB values</li> </ul> |
| | <ul> <li>N1 = patients with nonmissing values at both baseline and the specified</li> </ul> |
| | postbaseline analysis visit |
| Responder | Categorical descriptives for responders and nonresponders |
| | <ul> <li>N1 = patients with nonmissing values at both baseline and the specified</li> </ul> |
| | postbaseline analysis visit |

CFB = change from baseline

Two treatment cycles are defined in this analysis plan. Treatment Cycle 1 includes all visits from study baseline (also called cycle 1 baseline) to Week 24 or Exit visit if a patient receives throughout the study, or to the last visit before retreatment if a patient receives during the study. For visits in treatment Cycle 1, refer to study windows in Section 6.2. Treatment Cycle 2 applies to patients who receive retreatment, and includes all visits from retreatment and thereafter. Visits in treatment Cycle 2 will be determined based on the study days relative to the retreatment visit using the study windows specified in Section 6.2.

The study baseline value of an assessment will be the measurement prior to the treatment at Day 1 unless it is missing. In that case, the last nonmissing value recorded prior to the treatment (Day 1) will be used instead. The cycle baseline (also called cycle 2 baseline) value of an assessment will be the measurement prior to the retreatment at Week 12 from the first treatment unless it is missing. In that case, the last nonmissing value recorded prior to the retreatment (Week 12) will be used instead.

Ocular evaluation will be summarized by study eye and contralateral eye separately.

Some raw and derived data listings will be provided, and will be fully defined in the table, figure, and data listing specification document.

## **5.1.1.1.4 Missing Data**

General missing data handling conventions are summarized as follows:

- Missing data will not be imputed and all analyses will be based on observed data.
- Partial dates handling conventions are specified in Section 6.3, but will be listed in the data listings as they appear on the electronic case report forms (eCRFs).

## 5.1.1.2 Demographics

The safety population will be used to summarize demographics.

## 5.1.1.2.1 Analysis Populations

The distribution of patients within the analysis populations will be summarized as described in Table 5-3.

Table 5-3 Analysis Population Summaries

| Population | Description | Timing | Methodology |
|---|---|---|---|
| mITT and safety | Distribution in total and by treatment | | Categorical counts |
| populations | group | | |

## 5.1.1.2.2 Patient Disposition

Patient disposition encompasses the distribution of patients who enter, complete, and discontinue each specified analysis period, along with eCRF-reported discontinuation reasons from each respective analysis period. Patient disposition will be summarized as shown in Table 5-4.

Table 5-4 Patient Disposition Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Study disposition | Distribution in total and by treatment | During study | Categorical |
| | group | | descriptives |
| Patient disposition <sup>a</sup> by | Distribution in the safety population in | Treatment Period | Categorical |
| phase | total and by treatment group | | descriptives |

<sup>&</sup>lt;sup>a</sup> Patients who prematurely discontinued will be listed.

#### 5.1.1.2.3 Protocol Deviations

Protocol deviations will be defined in a separate document, including importance classification. Protocol deviations will be summarized as shown in Table 5-5.

Table 5-5 Protocol Deviation Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Significant protocol | Distribution in the safety population in | _ | Categorical |
| deviations <sup>a</sup> | total and by treatment group | | descriptives |

<sup>&</sup>lt;sup>a</sup> Patients with significant protocol deviations will be listed.

## 5.1.1.2.4 Demographics

Demographics will be summarized in total and by treatment group for the safety population as shown in Table 5-6.

Table 5-6 Demographic Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Age <sup>a</sup> | Age (years) relative to informed consent date | Informed consent | Continuous descriptives |
| Age group | <ul><li>&lt; 45 years</li><li>45-65 years</li><li>&gt; 65 years</li></ul> | Informed consent | Categorical descriptives |
| Sex, and race <sup>1</sup> | <ul> <li>eCRF categories</li> <li>Race group 1 <ul> <li>Caucasian</li> <li>Black</li> <li>Asian</li> <li>Hispanic</li> <li>Other</li> </ul> </li> <li>Race group 2 <ul> <li>Caucasian</li> <li>Non-caucasian</li> </ul> </li> </ul> | Screening period | Categorical<br>descriptives |

<sup>&</sup>lt;sup>a</sup> Patient demographics will be listed.

## 5.1.1.2.5 Medical History

Medical and ophthalmic history, encompassing abnormalities and surgeries reported as occurring before the Screening Visit, will be coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 19.0 or newer. Unique patients who report medical history events will be summarized by MedDRA system organ class (SOC) and preferred term (PT) in total and by treatment group for the safety population as shown in Table 5-7.

Table 5-7 Medical History Summary

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Medical history | Abnormalities and surgeries | Past | Categorical descriptives |
| Medical condition at trial initiation | Abnormalities and surgeries | Currently at the time informed consent was obtained | Categorical descriptives |
| Ophthalmic history | Ophthalmic abnormalities and surgeries | Past | Categorical descriptives |
| Ophthalmic condition at | Ophthalmic abnormalities and surgeries | Currently at the time | Categorical |

| Parameter | Description | Timing | Methodology |
|-----------------|-------------|------------------|--------------|
| trial nitiation | | informed consent | descriptives |
| | | was obtained | |

#### **5.1.1.2.6** Prior and Concomitant Medications

Medications will be coded using the WHO Drug Dictionary Enhanced (DDE), version MAR2016 or newer. Unique patients who reported medications will be summarized by MedDRA SOC, and PT, and WHO DDE drug base preferred name in total and by treatment group for the safety population as shown in Table 5-8.

**Table 5-8 Medication Summaries** 

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Prior medications | Medications taken ≥ 1 time before the study treatment start date, regardless of medication end date | Screening period | Categorical descriptives |
| Concomitant medications | Medications taken ≥ 1 time on or after the study treatment start date, regardless of medication start date | Treatment period | Categorical descriptives |

## **5.1.1.3** Exploratory Efficacy Analyses

## 5.1.1.3.1 Schirmer's Tear Test (With Anesthesia)

Schirmer's tear test (with anesthesia) will be summarized by treatment group as shown in Table 5-9.

Table 5-9 Schirmer's Tear Test Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Schirmer's tear test | Summary by analysis visit | Cycle 1: Study | CFB descriptives |
| score <sup>a</sup> | | baseline (Day 1) and | |
| | | Weeks 4, 8, 12, and | |
| | | 24 | |
| | | Cycle 2: Cycle<br>baseline and<br>Weeks 4R, 8R, and<br>12R | |
| Number (percent) of | Summary by analysis visit | Cycle 1: Weeks 4, 8, | Categorical |
| responders | • Responder defined as ≥ 10 mm/5 min | 12, and 24 | descriptives |
| | increase from study baseline in | | |
| | Schirmer's tear test score | | |

<sup>&</sup>lt;sup>a</sup> All schirmer's tear test data will be listed.

## 5.1.1.3.2 Tear Film Break-Up Time

Tear film break-up time (TBUT) will be summarized by treatment group as shown in Table 5-10.

Table 5-10 Tear Film Break-Up Time Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| TBUT | Summary by analysis visit | Cycle 1: Study | CFB descriptives |
| | • The average value of 3 measurements | baseline (Day 1) and | |
| | in each eye at each visit will be used | Weeks 4, 8, 12, and | |
| | | 24 | |
| | | Cycle 2: Cycle | |
| | | baseline and | |
| | | Weeks 4R, 8R, and | |
| | | 12R | |

## 5.1.1.3.3 Sodium Fluorescein Corneal Staining

Sodium fluorescein corneal staining will be summarized by treatment group as shown in Table 5-11.

Table 5-11 Sodium Fluorescein Corneal Staining Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| CFB in ordinal scale | Summary by analysis visit | Cycle 1: Study<br>baseline (Day 1) and<br>Weeks 4, 8, 12, and | CFB descriptives |
| | | Cycle 2: Cycle<br>baseline and<br>Weeks 4R, 8R, and<br>12R | |

## 5.1.1.3.4 Lissamine Green Conjunctival Staining

Lissamine green conjunctival staining will be summarized by treatment group as shown in Table 5-12.

Table 5-12 Lissamine Green Conjunctival Staining Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| CFB in ordinal scale of | Summary by analysis visit and by area | Cycle 1: Study | CFB descriptives |
| conjunctival staining | (nasal, temporal) and in total | baseline (Day 1) and | |
| | • Total is calculated as the sum of areas – | Weeks 4, 8, 12, and | |
| | nasal and temporal | 24 | |
| | | Cycle 2: Cycle | |
| | | baseline and | |
| | | Weeks 4R, 8R, and | |
| | | 12R | |

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| CFB in ordinal scale of total corneal and conjunctival staining | <ul> <li>Summary by analysis visit</li> <li>Total corneal and conjunctival staining is the sum of corneal staining plus conjunctival staining (nasal plus temporal)</li> </ul> | Cycle 1: Study<br>baseline (Day 1) and<br>Weeks 4, 8, 12, and<br>24 | CFB descriptives |
| | | Cycle 2: Cycle<br>baseline and<br>Weeks 4R, 8R, and<br>12R | |

## **5.1.1.3.5** Patient Symptoms (Visual Analog Scale)

A short questionnaire utilizing a VAS to quantify the severity of symptoms of dry eye will be administered. The questions refer to TODAY only including overall ocular discomfort from dry eye disease, level of discomfort experienced from symptoms as specified in Table 6-18. The score will be 0 to 100 with 0 = none and 100 = extreme.

Patient symptoms (VAS) will be summarized by treatment group as shown in Table 5-13.

Table 5-13 Patient Symptoms (Visual Analog Scale) Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Overall VAS score <sup>a</sup> | Summary by analysis visit | Cycle 1: Study | CFB descriptives |
| | | baseline (Day 1) and | |
| | | Weeks 12 and 24 | |
| | | Cyala 2: Cyala | |
| | | Cycle 2: Cycle | |
| | | baseline and | |
| | | Weeks 8R and 12R | |
| Worse VAS score <sup>a</sup> | Summary by analysis visit | Cycle 1: Study | CFB descriptives |
| | For each patient, the symptom among | baseline (Day 1) and | |
| | all 9 symptoms (specified in Table | Weeks 12 and 24 | |
| | 6-18) with the worst VAS at baseline | | |
| | (Day 1) will be used. If no single | Cycle 2: Cycle | |
| | symptom can be identified at baseline | baseline and | |
| | (Day 1), the symptom with the worst | Weeks 8R and 12R | |
| 2 | VAS score at screening will be used. | | |

<sup>&</sup>lt;sup>a</sup> All patient symptoms (VAS) data will be listed.

#### 5.1.1.3.6 Ocular Surface Disease Index

The Ocular Surface Disease Index (OSDI) Questionnaire consists of 12 questions based on which the total score (questions 1-12) and 3 subscales including ocular symptoms (questions 1-3), vision-related functioning (questions 4-9), and environmental triggers (questions 10-12) will be computed. The patients will be asked to rate each symptom using a 5-point scale (0 to 4), where 0 = none of the time, 1 = some of the time, 2 = half of the time, 3 = most of the time, and 4 = all of the time. Seven questions allow a response of not applicable (N/A). A higher score represents greater disability.

The OSDI Questionnaire scores will be summarized by treatment group as shown in Table 5-14.

Table 5-14 Ocular Surface Disease Index Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| OSDI score <sup>a</sup> | Summary by analysis visit and by | Cycle 1: Study | CFB descriptives |
| | <ul> <li>The total OSDI score</li> </ul> | baseline (Day 1) and | |
| | • The 3 subscale scores (specified in Table 6-20) | Weeks 4, 12, and 24 | |
| | , | Cycle 2: Cycle | |
| | | baseline and | |
| | | Weeks 4R and | |
| | | Week 12R | |
| Number (percent) of | Summary by analysis visit | Cycle 1: Weeks 4, | Categorical |
| responders | • Responder is defined as $\geq 20$ point | 12, and 24 | descriptives |
| | decrease from study baseline in total | | |
| | OSDI score | | |

<sup>&</sup>lt;sup>a</sup> All ocular surface disease index data will be listed.

## 5.1.1.3.7 Treatment Assessment by Investigator

The follow-up investigator will complete a global evaluation of the overall effect of investigational medication administered in reference to the Baseline visit (Day 1) prior to the of the investigational medication for each eye at the scheduled visits. The global evaluation score will be assessed based on the following scale:

- 0 = Completely cleared, no sign or symptom of disease
- 1 = Almost cleared: very significant clearance in disease with only traces of active disease remaining (approximately 90% improvement)
- 2 = Marked response: significant improvement with some disease remaining (approximately 75% improvement)
- 3 = Moderate response: intermediate improvement, between slight and marked (approximately 50% improvement)
- 4 = Slight response: some improvement in disease state but significant disease remains (approximately 25% improvement)
- 5 = Condition unchanged
- 6 = Condition worsened

Treatment assessment by investigator will be summarized by treatment group as shown in Table 5-15.

Table 5-15 Treatment Assessment by Investigator Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Global evaluation | Summary by analysis visit for the raw score | Cycle 1: Weeks 8, | Continuous |
| score | | 12, and 24 | descriptives |
| | | Cycle 2: Week 8R, | |
| | | and Week 12R | |

## **5.1.1.4** Safety Analyses

Safety analyses will be based on the safety population.

## **5.1.1.4.1 Study Treatment Exposure**

Study treatment exposure and compliance will be summarized by treatment group for the safety population as shown in Table 5-16.

Table 5-16 Study Treatment Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Study treatment | Date of study exit – date of 1st injection + 1 | Treatment period | Continuous |
| exposure (days) | | | descriptives |

#### 5.1.1.4.2 Adverse Events

Adverse events (AEs) are defined as shown in Table 5-17.

Table 5-17 AE Terms

| Term | Description |
|---|---|
| TEAE | An adverse event recorded on the eCRF would be considered treatment-emergent if either of |
| | the following conditions are met: |
| | AE onset date ≥ first study treatment date; or |
| | AE onset date < first study treatment date and either: |
| | the severity of the event worsened on or after the first study treatment date, or |
| | the event became serious on or after the first study treatment date |
| SeriousTEAE | An event identified as TEAE that further meets SAE criteria at any time would be a serious |
| | TEAE. |

SAE = serious adverse event; TEAE = treatment-emergent adverse event

AEs, encompassing abnormalities and surgeries reported as occurring after the Screening Visit, will be coded using MedDRA version 19.0 or newer. Unique patients reporting AEs in the following AE categories will be summarized by treatment group for the safety population as shown in Table 5-18.

Table 5-18 AE Summaries

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| Overall summary | Overall summary for the following | From treatment start | Categorical |
| | categories: | date until | descriptives |
| | <ul> <li>TEAEs (ocular vs. non-ocular)</li> </ul> | Week 24/Week 12R or | |
| | Study drug-related TEAEs (ocular vs. non-ocular) Study drug-related TEAEs | early termination date,<br>whichever comes first | |
| | • Study procedure-related TEAEs (ocular vs. non-ocular) | | |
| | <ul> <li>Serious TEAEs (ocular vs. non-<br/>ocular)</li> </ul> | | |
| | <ul> <li>TEAEs leading to study</li> </ul> | | |

| Parameter | Description | Timing | Methodology |
|---|---|---|---|
| | discontinuation (ocular vs. non- | | |
| | ocular) | | |
| | • Deaths | | |
| TEAEs <sup>a</sup> | Overall summary and by SOC in | From treatment start | Categorical |
| | alphabetical order, PT and worst severity | date until | descriptives |
| | The worst severity is defined as the greater | Week 24/Week 12R | |
| | The worst severity is defined as the greater of the onset severity and maximum | or early termination date, whichever comes | |
| | severity following onset recorded on the | first | |
| | eCRF. If the same TEAE term has been | IIISt | |
| | reported more than once for a subject with | | |
| | different severity grades, the worst severity | | |
| | grade will be used in the tabulation. | | |
| Ocular TEAEs | Overall summary and by SOC in | From treatment start | Categorical |
| | alphabetical order, PT and worst severity | date until | descriptives |
| | | Week 24/Week 12R | |
| | The worst severity is defined as the greater | or early termination | |
| | of the onset severity and maximum | date, whichever comes | |
| | severity following onset recorded on the | first | |
| | eCRF. If the same TEAE term has been | | |
| | reported more than once for a subject with | | |
| | different severity grades, the worst severity grade will be used in the tabulation. | | |
| Study drug-related | Overall summary and by SOC in | From treatment start | Categorical |
| ocular TEAEs | alphabetical order and PT | date until | descriptives |
| Oddiai TEITES | aipinaoettear oraer ana 1 1 | Week 24/Week 12R | descriptives |
| | | or early termination | |
| | | date, whichever comes | |
| | | first | |
| Study procedure-related | Overall summary and by SOC in | From treatment start | Categorical |
| ocular TEAEs | alphabetical order and PT | date until | descriptives |
| | | Week 24/Week 12R | |
| | | or early termination | |
| | | date, whichever comes | |
| Serious TEAEs | Overall summers and by SOC in | first From treatment start | Categorical |
| SCHOUS LEAES | Overall summary and by SOC in alphabetical order and PT | date until | descriptives |
| | alphabetical order and 1 1 | Week 24/Week 12R | descriptives |
| | | or early termination | |
| | | date, whichever comes | |
| | | first | |
| TEAEs leading to study | Overall summary and by SOC in | From treatment start | Categorical |
| discontinuation | alphabetical order and PT | date until | descriptives |
| | | Week 24/Week 12R | |
| | | or early termination | |
| | | date, whichever comes | |
| | | first | |

eCRF = electronic case report form; PT = preferred term; SAE = serious adverse event; SOC = system organ class; TEAE = treatment-emergent adverse event

a All AEs including pretreatment AEs and TEAEs, and SAEs will be listed.

## **5.1.1.4.3** Clinical Laboratory Assessments

Clinical laboratory assessments will be summarized by treatment group for the safety population as shown in Table 5-19.

Table 5-19 Clinical Laboratory Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Descriptives | Summary by laboratory category, | Cycle 1: Study | CFB descriptives |
| | parameter and analysis visit | baseline (screening), | |
| | <ul> <li>Parameters specified in Table</li> </ul> | Week 12 (for | |
| | 6-22 | Cohorts 6C and 6D | |
| | | only), and Week 24 | |
| | | Cycle 2: Cycle | |
| | | baseline and | |
| | | Week 12R | |

## **5.1.1.4.4 Vital Signs**

Vital signs will be summarized by treatment group for the safety population as shown in Table 5-20.

Table 5-20 Vital Signs Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Descriptives | Summary by parameter and analysis visit | Cycle 1: Study | CFB descriptives |
| | <ul> <li>Parameters specified in Table</li> </ul> | baseline andWeeks | |
| | 6-23 | 1, 8, 12 (for Cohorts | |
| | | 6C and 6D only), | |
| | | and 24 | |
| | | Cycle 2: Cycle | |
| | | baseline, Day 1R, | |
| | | and Week 12R | |

## 5.1.1.4.5 Other Safety Analyses

## 5.1.1.4.5.1 Best-Corrected Visual Acuity

Manifest refraction will be performed at screening and used for BCVA at all subsequent visits until study exit. If there is a decrease in BCVA, the manifest refraction should be repeated as confirmation. Visual acuity (in Snellen equivalents) will be measured for each eye using a logarithmic visual acuity chart for testing at 10 feet (3 meters) at the scheduled visits.

The visual acuity will be recorded on the eCRF in Snellen equivalent units (eg, 20/63) as the lowest line read with 1 or 0 mistakes.

The line CFB at each evaluation is calculated using the following algorithm:

line change =  $(10)*[\log_{10} (XB/20) - \log_{10} (XF/20)]$ , where

- XB = denominator of the Snellen equivalent unit at baseline
- XF = denominator of the Snellen equivalent unit at post treatment visit

Each logarithmic value is to be rounded to the nearest tenth before subtraction. A positive value indicates an improvement and a negative value indicates a worsening. For example, the line change for a Snellen equivalent unit of 20/25 at baseline followed by a Snellen equivalent unit of 20/80 at day 2 would be

Line change = 
$$10 \times [\log_{10}(25/20) - \log_{10}(80/20)] = 10 \times (0.1 - 0.6) = -5$$

which represents a worsening of 5 lines in visual acuity.

BCVA will be summarized by treatment group for the safety population as shown in Table 5-21.

Table 5-21 BCVA Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Line CFB <sup>a</sup> | Summary by analysis visit and line change | Cycle 1: Day 2 and | Categorical |
| | categories defined below or line change of | Weeks 1, 2, 4, 8, 12, | descriptives |
| | $\leq -2, -1, 0, +1, \text{ or } \geq +2$ : | and 24 | |
| | • Better (line changes of $\geq +2$ ) | | |
| | • No change (line changes of -1, 0, | Cycle 2: Day 1R | |
| | +1) | and Weeks 1R, 4R, | |
| | ○ Line change of +1 | 8R, and 12R | |
| | o Line change of 0 | | |
| | o Line change of -1 | | |
| | • Worse (line changes of $\leq$ -2) | | |

CFB = change from baseline

## 5.1.1.4.5.2 Macroscopic Bulbar Hyperemia

The macroscopic (gross) bulbar hyperemia grading consists of global assessments and regional assessments, which will be done under consistent illumination by comparing the appearance of the bulbar conjunctiva to standard photographs (Allergan bulbar conjunctival hyperemia grading guide) at the scheduled visits. Regional assessment includes superior temporal, superior nasal, inferior temporal, and inferior nasal assessment. It will be graded using a 5-point scale described as follows:

```
0
       (None)
                          Normal: vessels of bulbar conjunctiva easily observed
+0.5
       (Trace)
                    =
                          Trace flush, reddish-pink color
                         Mild flush, reddish color
+1
       (Mild)
       (Moderate)
                          Bright red color
+2
                    =
                         Deep, bright diffuse redness
+3
       (Severe)
```

<sup>&</sup>lt;sup>a</sup> All BCVA will be listed.

Macroscopic bulbar hyperemia will be summarized by treatment group for the safety population as shown in Table 5-22.

Table 5-22 Macroscopic Bulbar Hyperemia Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Global assessment: | Summary by analysis visit | Cycle 1: Study | Categorical |
| severity grade | | baseline (Day 1), | descriptives |
| | | Day 2, and Weeks 1, | |
| | | 2, 4, 8, 12, and 24 | |
| | | Cycle 2: Cycle | |
| | | baseline, Day 1R, | |
| | | and Weeks 1R, 4R, | |
| | | 8R, and 12R | |

## 5.1.1.4.5.3 Slit-lamp Biomicroscopy

Slit-lamp biomicroscopy will be summarized by treatment group for the safety population. Biomicroscopy findings will be coded using MedDRA terminology and summarized for each eye by treatment group as shown in Table 5-23.

Table 5-23 Slit-lamp Biomicroscopy Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| One or more severity | Overall summary and by PT | From treatment start | Categorical |
| grade increase from | | date until | descriptives |
| baseline | | Week 24/Week 12R | _ |
| | | or early termination | |
| | | date, whichever | |
| | | comes first | |

PT = preferred term

## **5.1.1.4.5.4 Dilated Ophthalmic Examinations**

Ophthalmoscopy findings will be coded using MedDRA terminology.

Cup/disc ratio will be reported using a 0.0 to 1.0 scale. The Armaly chart provided by Allergan provides a pictorial scale of cup/disc ratio of 0.0 to 0.8. Only listing will be provided for cup/disc ratio.

Dilated ophthalmic examinations will be summarized by treatment group for the safety population as shown in Table 5-24.

Table 5-24 Dilated Ophthalmic Examinations Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| One or more severity | Overall summary and by PT | Week 12 (for | Categorical |
| grade increase from | | Cohorts 6C and 6D | descriptives |
| baseline | | only), | _ |
| | | Week 24/Week 12R | |
| | | or early termination | |
| | | date, whichever | |
| | | comes first | |

PT = preferred term

## 5.1.1.4.5.5 Photographic Conjunctival Hyperemia

The photographic conjunctival hyperemia grading consists of global assessments and regional assessments, which will be done using a Canfield camera in each eye at the scheduled visits. Global assessment includes global, global nasal and global temporal assessment, and regional assessment includes superior temporal, superior nasal, inferior temporal, and inferior nasal assessment. It will be graded as 0 = none, +0.5 = trace, +1 = mild, +2 = moderate, +3 = severe, +3 = connot grade, and +3 = connot grade, and +3 = connot grade, and +3 = connot grade.

Photographic conjunctival hyperemia will be summarized by treatment group for the safety population as shown in Table 5-25.

Table 5-25 Photographic Conjunctival Hyperemia Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Global assessment: | Summary by analysis visit | Cycle 1: Study | Categorical |
| severity grade | | baseline (Day 1), | descriptives |
| | | Day 2, and Weeks 1, | |
| | | 2, 4, 8, 12, and 24 | |
| | | Cycle 2: Cycle | |
| | | baseline, Day 1R, | |
| | | and Weeks 1R, 4R, | |
| | | 8R, and 12R | |

#### 5.1.1.4.5.6 Intraocular Pressure

Measurement of intraocular pressure (IOP) will be taken for each eye using the Goldmann applanation tonometer affixed to a slit lamp at the scheduled visits.

IOP will be summarized by treatment group for the safety population as shown in Table 5-26.

Table 5-26 Intraocular Pressure Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| IOP <sup>a</sup> | Summary by analysis visit | Cycle 1: Study | CFB descriptives |
| | | baseline (Day 1), | |
| | | Week 12 (for | |
| | | Cohorts 6C and 6D | |
| | | only), and Week 24 | |
| | | Cycle 2: Cycle | |
| | | baseline, Week 12R | |

IOP = intraocular pressure

## **5.1.1.4.5.7 REFRESH PLUS Use**

REFRESH PLUS use will be summarized by treatment group for the safety population as shown in Table 5-27.

Table 5-27 REFRESH PLUS Use and Compliance Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| REFRESH PLUS descriptives | Summary by analysis visit | Cycle 1: Study baseline (Day 1), Day 2, and Weeks 1, | CFB descriptives |
| | | 2, 4, 8, 12, and 24 Cycle 2: Cycle baseline, Day 1R, and Weeks 1R, 4R, 8R, and 12R | |

## **5.1.1.5** Health Outcomes Data Analyses

The Supplemental Dry Eye Patient Reported Outcomes Questionnaire is a series of questions designed to gather information about the types and severity of dry eye symptoms that are experienced by patients in each eye. Health outcomes data will be summarized by treatment group for the mITT Population as shown in Table 5-28.

Table 5-28 Health Outcomes Data Summaries

| Endpoint | Description | Timing | Methodology |
|---|---|---|---|
| Treatment satisfaction | Summary of raw score by analysis visit | Cycle 1: Weeks 4, 8, | Continuous |
| | | 12, and 24 | descriptives |

<sup>&</sup>lt;sup>a</sup> All IOP data will be listed.

| Endpoint | Description | Timing | Methodology |
|----------|-------------|--------------------|-------------|
| | | Cycle 2: Weeks 4R, | |
| | | 8R, and 12R | |

## 5.1.1.6 Subgroup Analyses

Subgroup analyses are not planned for stage 1.

## 5.1.1.7 Interim Analyses

An interim database lock of stage 1 will not be conducted until after all patients in Cohorts 1 through 6B complete the study and all patients in Cohorts 6C and 6D complete at least Week 1 following retreatment. Statistical analyses will be performed following the database lock to support the design of future clinical studies.

## **5.1.2 Determination of Sample Size**

The sample size for stage 1 is determined empirically.

<u>Stage 1</u>: Stage 1 will have up to 63 patients and approximately 10 cohorts (Cohorts 1 to 6D). The anticipated numbers of patients per cohort are 3 for Cohort 1; 4 each for Cohorts 2, 6C, and 6D; and 8 each for Cohorts 3 through 6B.

## **5.2** Changes in the Conduct of the Study or Planned Analyses

## 5.2.1 Changes in the Conduct of the Study

Not applicable.

## **5.2.2** Changes to Analyses Prior to Database Lock

The definition of modified intent-to-treat (mITT) population is changed to all randomized patients who have baseline and at least 1 postbaseline assessment for 1 or more of the exploratory efficacy measurements from all patients who receive study treatment and have baseline and at least 1 postbaseline assessment for 1 or more of the exploratory efficacy measurements.

# 6. Data Handling and Analysis Conventions

## 6.1 Study Treatment Conventions

## 6.1.1 Analysis Days

Treatment days are defined as shown in Table 6-1.

Table 6-1 Analysis Day Definitions

| Term | Description |
|---|---|
| Treatment Day | Relative to treatment start date |
| | If analysis date ≥ treatment start date: |
| | • Day = analysis date – treatment start date + 1 |
| | <ul> <li>Day 1 = treatment start date</li> </ul> |
| | If analysis date < treatment start date: |
| | • Day = analysis date – treatment start date |
| | <ul> <li>Day -1 = day before treatment start date</li> </ul> |
| | o There is no Day 0 |

## 6.2 Analysis Visit Windows

All stage 1 analyses will be performed based on the analysis visit windows defined below.

The analysis visit windows for exploratory efficacy and safety endpoints follow the schedule of visits in the protocol and are defined as follows:

## **6.2.1** Treatment Cycle 1

Table 6-2 Analysis Visit Definitions 1

| Analysis Phase | Analysis Visit<br>(Derived) | Target Number of Days<br>from Treatment | Window <sup>a</sup> |
|---|---|---|---|
| Pretreatment | Study Baseline | Day 1 | Treatment Day 1 |
| Treatment | Day 2 | Day 2 | Treatment Day [2, 4] |
| | Week 1 | Day 7 | Treatment Day [5, 10] |
| | Week 2 | Day 14 | Treatment Day [11, 20] |
| | Week 4 | Day 28 | Treatment Day [21, 41] |
| | Week 8 | Day 56 | Treatment Day [42, 69] |
| | Week 12 | Day 84 | Treatment Day [70, 125] |
| | Week 24 | Day 168 | Treatment Day ≥126 |

For endpoints with scheduled visits of Study Baseline (Day 1), Day 2, Week 1, Week 2, Week 4, Week 8, Week 12, and Week 24

Table 6-3 Analysis Visit Definitions 2

| Analysis Phase | Analysis Visit<br>(Derived) | Target Number of Days from Treatment | Window <sup>a</sup> |
|---|---|---|---|
| Pretreatment | Study Baseline | Day 1 | Treatment Day 1 |
| Treatment | Week 4 | Day 28 | Treatment Day [2, 41] |

<sup>&</sup>lt;sup>a</sup> Study days are calculated based on the visit date – Treatment (Day 1) visit date + 1.

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Treatment | Window <sup>a</sup> |
| | Week 8 | Day 56 | Treatment Day [42, 69] |
| | Week 12 | Day 84 | Treatment Day [70, 125] |
| | Week 24 | Day 168 | Treatment Day >=126 |

For endpoints with scheduled visits of Study Baseline (Day 1), Week 4, Week 8, Week 12, and Week 24.

Table 6-4 Analysis Visit Definitions 3

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Treatment | Window <sup>a</sup> |
| Pretreatment | Study Baseline | Day 1 | Treatment Day 1 |
| | Week 1 | Day 7 | Treatment Day [2, 31] |
| T | Week 8 | Day 56 | Treatment Day [32, 69] |
| Treatment | Week 12 | Day 84 | Treatment Day [70, 125] |
| | Week 24 | Day 168 | Treatment Day >=126 |

For endpoints with scheduled visits of Study Baseline (Day 1), Week 1, Week 8, Week 12, and Week 24.

Table 6-5 Analysis Visit Definitions 4

| Analysis Phase | Analysis Visit<br>(Derived) | Target Number of Days from Treatment | Window <sup>a</sup> |
|---|---|---|---|
| Pretreatment | Study Baseline | Day 1 | Treatment Day 1 |
| | Week 1 | Day 7 | Treatment Day [2, 31] |
| Treatment | Week 8 | Day 56 | Treatment Day [32, 111] |
| | Week 24 | Day 168 | Treatment Day >=112 |

For endpoints with scheduled visits of Study Baseline (Day 1), Week 1, Week 8, and Week 24.

Table 6-6 Analysis Visit Definitions 5

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Treatment | Window <sup>a</sup> |
| Pretreatment | Study Baseline | Day 1 | Treatment Day 1 |
| | Week 4 | Day 28 | Treatment Day [2, 55] |
| Treatment | Week 12 | Day 84 | Treatment Day [56, 125] |
| | Week 24 | Day 168 | Treatment Day >=126 |

For endpoints with scheduled visits of Study Baseline (Day 1), Week 4, Week 12, and Week 24.

<sup>&</sup>lt;sup>a</sup> Study days are calculated based on the visit date – Treatment (Day 1) visit date + 1.

Table 6-7 Analysis Visit Definitions 6

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Treatment | Window <sup>a</sup> |
| | Week 8 | Day 56 | Treatment Day [2, 69] |
| Treatment | Week 12 | Day 84 | Treatment Day [70, 125] |
| | Week 24 | Day 168 | Treatment Day >=126 |

For endpoints with scheduled visits of Week 8, Week 12, and Week 24.

Table 6-8 Analysis Visit Definitions 7

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| Analysis Phase | (Derived) | from Treatment | Window <sup>a</sup> |
| Pretreatment | Study Baseline | Day 1 | Treatment Day 1 |
| Treatment | Week 12 | Day 84 | Treatment Day [2, 125] |
| | Week 24 | Day 168 | Treatment Day >=126 |

For endpoints with scheduled visits of Study Baseline (Day 1), Week 12, and Week 24.

Table 6-9 Analysis Visit Definitions 8

| Analysis Phase | Analysis Visit (Derived) | Target Number of Days from Treatment | Window <sup>a</sup> |
|---|---|---|---|
| Pretreatment | Study Baseline | Day 1 | Treatment Day 1 |
| Treatment | Week 24 | Day 168 | Treatment Day >=2 |

For endpoints with scheduled visits of Study Baseline (Day 1), and Week 24.

## **6.2.2** Treatment Cycle 2

Table 6-10 Analysis Visit Definitions 1 (Retreatment)

| | Analysis Visit<br>(Derived) | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | , | from Retreatment | Window <sup>a</sup> |
| Pre-retreatment | Cycle Baseline | Day 1 | Retreatment Day 1 (Week 12 from |
| | | | treatment start) |
| | Day 1R | Day 2 | Treatment Day [2, 4] |
| Datasatusant | Week 1R | Day 7 | Treatment Day [5, 17] |
| Retreatment | Week 4R | Day 28 | Treatment Day [18, 41] |
| | Week 8R | Day 56 | Treatment Day [42, 69] |
| | Week 12R | Day 84 | Treatment Day ≥70 |

For endpoints with scheduled visits of Cycle Baseline (Day 1), Day 1R, Week 1R, Week 4R, Week 8R, and Week 12R.

<sup>&</sup>lt;sup>a</sup> Study days are calculated based on the visit date – Treatment (Day 1) visit date + 1.

<sup>&</sup>lt;sup>a</sup> Study days are calculated based on the visit date – Treatment (Day 1) visit date + 1.

<sup>&</sup>lt;sup>a</sup> Study days are calculated based on the visit date – Treatment (Day 1) visit date + 1.

<sup>&</sup>lt;sup>a</sup> Study days from retreatment are calculated based on the visit date – retreatment visit date + 1.

Table 6-11 Analysis Visit Definitions 2 (Retreatment)

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Retreatment | Window <sup>a</sup> |
| Pre retreatment | Cycle Baseline | Day 1 | Retreatment Day 1 (Week 12 from |
| | | | treatment start) |
| | Week 4R | Day 28 | Treatment Day [2, 41] |
| Retreatment | Week 8R | Day 56 | Treatment Day [42, 69] |
| | Week 12R | Day 84 | Treatment Day ≥ 70 |

For endpoints with scheduled visits of Cycle Baseline (Day 1), Week 4R, Week 8R, and Week 12R.

Table 6-12 Analysis Visit Definitions 3 (Retreatment)

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Retreatment | Window <sup>a</sup> |
| Pre retreatment | Cycle Baseline | Day 1 | Retreatment Day 1 (Week 12 from treatment start) |
| Datusatusant | Day 1R | Day 2 | Treatment Day [2, 42] |
| Retreatment | Week 12R | Day 84 | Treatment Day $\geq 43$ |

For endpoints with scheduled visits of Cycle Baseline (Day 1), Day 1R, and Week 12R.

Table 6-13 Analysis Visit Definitions 4 (Retreatment)

| Analysis Phase | Analysis Visit<br>(Derived) | Target Number of Days from Retreatment | Window <sup>a</sup> |
|---|---|---|---|
| Pre retreatment | Cycle Baseline | Day 1 | Retreatment Day 1 (Week 12 from |
| | | | treatment start) |
| D - 4 4 4 | Week 8R | Day 56 | Treatment Day [2, 69] |
| Retreatment | Week 12R | Day 84 | Treatment Day ≥ 70 |

For endpoints with scheduled visits of Cycle Baseline (Day 1), Week 8R, and Week 12R.

Table 6-14 Analysis Visit Definitions 5 (Retreatment)

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Retreatment | Window <sup>a</sup> |
| Pre retreatment | Cycle Baseline | Day 1 | Retreatment Day 1 (Week 12 from treatment start) |
| Datasatusant | Week 4R | Day 28 | Treatment Day [2, 55] |
| Retreatment | Week 12R | Day 84 | Treatment Day $\geq 56$ |

For endpoints with scheduled visits of Cycle Baseline (Day 1), Week 4R, and Week 12R.

<sup>&</sup>lt;sup>a</sup> Study days from retreatment are calculated based on the visit date – retreatment visit date + 1.

Table 6-15 Analysis Visit Definitions 6 (Retreatment)

| | Analysis Visit | Target Number of Days | |
|---|---|---|---|
| <b>Analysis Phase</b> | (Derived) | from Retreatment | Window <sup>a</sup> |
| Pre retreatment | Cycle Baseline | Day 1 | Retreatment Day 1 (Week 12 from |
| | | | treatment start) |
| Retreatment | Week 12R | Day 84 | Treatment Day $\geq 2$ |

For endpoints with scheduled visits of Cycle Baseline (Day 1), and Week 12R.

The following general conventions will apply unless otherwise specified:

- If both scheduled and unscheduled visits occur within a single window, the scheduled visit will be used; unscheduled visits will be used only if there is no scheduled visits available in that window. If multiple visits are eligible for windowing within a single visit window, the visit closest to the target day will be used in the analysis. If multiple visits are equidistant to the target day, the latest visit will be used.
- For clinical laboratory variables, the latest nonmissing assessment within any analysis window will be flagged as the analysis value. This rule will be applied separately for each variable for nonmissing data only. (The exception is because re–runs of laboratory variables may only involve one or a few variables and would thus include missing data for many variables)
- All assessments will be included in respective listings.

## 6.3 Missing/Incomplete Date Conventions

Dates may be imputed with year, month, and day values under certain scenarios:

**Table 6-16 Imputation Scenarios** 

| | | Complete | | |
|----------|------|----------|-----|-----------------|
| Scenario | Year | Month | Day | Imputable |
| 1 | Yes | Yes | Yes | Complete |
| 2 | Yes | Yes | | Yes |
| 3 | Yes | _ | Yes | No <sup>a</sup> |
| 4 | Yes | _ | | Yes |
| 5 | _ | Yes | Yes | No <sup>a</sup> |
| 6 | _ | Yes | | No <sup>a</sup> |
| 7 | _ | _ | Yes | No <sup>a</sup> |
| 8 | _ | _ | _ | Yes |

<sup>&</sup>lt;sup>a</sup> Not allowed per database design.

Dates will be imputed initially toward a specified target date for imputable scenarios 2, 4, and 8, and adjusted against the latest reasonable dates. The initial imputed date is determined by the algorithm show in Table 6-17.

<sup>&</sup>lt;sup>a</sup> Study days from retreatment are calculated based on the visit date – retreatment visit date + 1.

Table 6-17 Initial Imputed Date Algorithm

| Available Year | | Available Month (MM) | | |
|---|---|---|---|---|
| (YYYY) | Missing | < Target Month | = Target Month | > Target Month |
| Missing | Target Date | | _ | |
| < Target Year | YYYY-12-31 | | YYYY-MM-LD | |
| = Target Year | Target Date | YYYY-MM-LD | Target Date | YYYY-MM-01 |
| > Target Year | YYYY-01-01 | | YYYY-MM-01 | |

YYYY = available start date year; MM = available start date month; LD = last day of the month.

## 6.3.1 Missing/Incomplete AE Start Date

AE start dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = treatment start date
- Complete end date

## 6.3.2 Missing/Incomplete Medication Start Date

Medication start dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = treatment start date -1
- Complete end date

## 6.3.3 Missing/Incomplete AE/Medication End Date

AE and medication end dates will be imputed as the minimum of the following:

- Initial imputed date, where target date = from treatment start date until Week 24/Week 12R or early termination date, whichever comes first
- Death date





## 6.5 Safety Endpoint Conventions

## 6.5.1 Adverse Events

## 6.5.1.1 Missing Intensity or Relationship

If the investigator is unable to provide the actual values, the imputations will be applied as shown in Table 6-21.

Table 6-21 Missing AE Intensity and Relationship Imputation Algorithms

| Missing Value | Imputation | Timing |
|---------------|--------------|------------------|
| Intensity | Mild | Screening Period |
| | Severe | Treatment Period |
| Relationship | <del>_</del> | Screening Period |
| l | Related | Treatment Period |

## 6.5.2 Clinical Laboratory Assessments

The laboratory parameters will be included as shown in Table 6-22.

Table 6-22 Clinical laboratory Parameters

| Category | Parameters |
|---|---|
| Hematology | Hematocrit, hemoglobin, HbA1c mean corpuscular hemoglobin (MCH), mean corpuscular |
| | hemoglobin concentration (MCHC), mean corpuscular volume (MCV), platelets, red blood cell |
| | (RBC) count, RBC morphology, total white blood cell (WBC) count, and differential (neutrophils, |
| | bands, lymphocytes, monocytes, basophils, and eosinophils) |
| Chemistry | Albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartase aminotransferase (AST), |
| | gamma-glutamyl transferase (GGT), bicarbonate, calcium, chloride, creatinine, creatine kinase, |
| | direct bilirubin, glucose, indirect bilirubin, magnesium, phosphorous, potassium, sodium, total |
| | bilirubin, total cholesterol, total protein, urea nitrogen, and uric acid |
| Urinalysis | Specific gravity, pH, color, protein, glucose, blood, bilirubin, and microscopic examination (WBC, |
| | RBC, epithelial cells, bacteria, mucus, casts, crystals) |

## 6.5.3 Vital Signs

The vital sign parameters as shown in Table 6-23 will be summarized.

Table 6-23 Vital Sign Descriptive Parameters

| Parameters | |
|---|---|
| Systolic blood pressure (mmHg) Diastolic blood pressure (mmHg) | Pulse rate (bpm) |

# 6.5.4 Slit-lamp Biomicroscopy

The slit-lamp biomicroscopy examination consists of evaluation of the eye area/condition using a 5-point or 6-point scales, as well as present no or yes, as shown in Table 6-24.

Table 6-24 Slit-lamp Biomicroscopy Scales

| Eye Area/Condition | | |
|---|---|---|
| Eyelids/Eyelid Margins/Lashes | 0 | (None) |
| • Edema (eyelids) | +0.5 | (Trace) |
| • Erythema | +1 | (Mild) |
| Conjunctiva (Bulbar or Palpebral) | +2 | (Moderate) |
| Hyperemia | +3 | (Severe) |
| • Edema | | |
| <ul> <li>Subconjunctival Hemorrhage</li> </ul> | | |
| Cornea | | |
| • Edema | | |
| Superficial Punctate Keratopathy | | |
| Anterior Chamber | 0 = | 0 cells |
| • Cells | +0.5 = | 1 to 5 cells (trace) |
| | +1 = | 6 to 15 cells |

| Eye Area/Condition | Scale |
|---|---|
| | +2 = 16 to 25 cells |
| | +3 = 26 to 50 cells |
| | +4 = > 50 cells |
| Anterior Chamber | 0 = None: no flare seen |
| • Flare | +1 = Faint: faint flare seen |
| | +2 = Moderate: iris and lens details clear |
| | +3 = Marked: iris and lens details hazy |
| | +4 = Intense: fibrin or plastic aqueous |
| Presence of Iris/Pupil Pathology and Other Pathology | Yes |
| | No |
| Other Pathology if present | +0.5 (trace) |
| | +1 (mild) |
| | +2 (moderate) |
| | +3 (severe) |

## Explanation:

## Eyelids/Eyelid Margins/Lashes

#### Edema (eyelids)

| 0 | (None) | No edema |
|------|------------|-------------------------------------|
| +0.5 | (Trace) | Localized, minimal (trace) swelling |
| +1 | (Mild) | Localized, mild swelling |
| +2 | (Moderate) | Diffuse, moderate swelling |
| +3 | (Severe) | Diffuse, severe swelling |

## Erythema

| 0 | (None) | No erythema |
|---|---|---|
| +0.5 | (Trace) | Localized, minimal (trace) flush reddish color |
| +1 | (Mild) | Localized, mild, flush reddish color |
| +2 | (Moderate) | Diffuse reddish color encompassing the entire lid margin |
| +3 | (Severe) | Deep diffuse reddish color of lid margins and superior and/or inferior eyelid |

## Conjunctiva (Bulbar or Palpebral)

## **Hyperemia**

| 0 | (None) | No hyperemia |
|------|------------|--------------------------------------|
| +0.5 | (Trace) | Minimal (trace) flush, reddish color |
| +1 | (Mild) | Mild flush, reddish color |
| +2 | (Moderate) | Bright red color |
| +3 | (Severe) | Deep, bright diffuse redness |

## <u>Edema</u>

| 0 | (None) | No edema |
|------|---------|-------------------------------------|
| +0.5 | (Trace) | Localized, minimal (trace) swelling |

| +1 | (Mild) | Localized, mild swelling |
|----|------------|----------------------------|
| +2 | (Moderate) | Diffuse, moderate swelling |
| +3 | (Severe) | Diffuse, severe swelling |

#### Subconjunctival Hemorrhage

| 0 | (None) | No hemorrhage |
|---|---|---|
| +0.5 | (Trace) | Flat hemorrhage ≤ 1 quadrant |
| +1 | (Mild) | Elevated hemorrhage $\leq 1$ quadrant, or flat and $\geq 1$ quadrant |
| +2 | (Moderate) | Elevated hemorrhage $> 1$ but $\le 2$ quadrants |
| +3 | (Severe) | Elevated hemorrhage > 2 quadrants |

#### Cornea

#### Edema

| Lucina | | |
|---|---|---|
| 0 | (None) | No edema |
| +0.5 | (Trace) | Localized, minimal (trace) epithelial haze |
| +1 | (Mild) | Dull glass appearance of epithelium that may include fine localized microcystic changes |
| +2 | (Moderate) | Dull glass appearance of epithelium with large number of cystic changes with or without |
| | | stromal edema |
| +3 | (Severe) | Epithelial bullae and/or stromal edema, localized or diffuse, with or without stromal |
| | | striae |

#### Superficial Punctate Keratopathy

| 0 | = | No superficial punctate keratopathy |
|------|---|-------------------------------------|
| +0.5 | = | Trace |
| +1 | = | Mild |
| +2 | = | Moderate |
| +3 | = | Severe |

#### **Anterior Chamber**

#### Cells

| 0 | = | 0 cells |
|------|---|----------------------|
| +0.5 | = | 1 to 5 cells (trace) |
| +1 | = | 6 to 15 cells |
| +2 | = | 16 to 25 cells |
| +3 | = | 26 to 50 cells |
| +4 | = | > 50 cells |

#### Flare 0

| +1 | = | Faint: faint flare seen |
|----|---|---------------------------------------|
| +2 | = | Moderate: iris and lens details clear |
| +3 | = | Marked: iris and lens details hazy |
| +4 | = | Intense: fibrin or plastic aqueous |

= None: no flare seen

## Iris/Pupil and Other Pathology

The presence of iris/pupil pathology and any other pathology will be evaluated. Other pathology will be graded as +0.5 = trace, +1 = mild, +2 = moderate, and +3 = severe.

## 6.5.5 Dilated Ophthalmic Examinations

The evaluation of dilated ophthalmic examinations is shown in Table 6-25.

Table 6-25 Dilated Ophthalmic Examinations Grade

| Description | | | Grade |
|---|---|---|---|
| Lens Status: | | Severity: | |
| <ul> <li>Phakic</li> </ul> | | 0 | (None) |
| 0 | Cortical lens opacity | 1 | (Mild) |
| 0 | Nuclear lens opacity | 2 | (Moderate) |
| 0 | Posterior Subcapsular lens opacity | 3 | (Severe) |
| <ul> <li>Pseudophakic</li> </ul> | | | |
| • Aphak | ic | | |
| Presence of Other Pathology | | Yes | |
| | | No | |
| Other pathology if present: | | +0.5 | (Trace) |
| • Lens | | +1 | (Mild) |
| Vitreou | ıs | +2 | (Moderate) |
| • Fundus | S | +3 | (Severe) |
| Optic nerve | | NE | (Not Evaluable) |

# **6.6** Health Outcomes Endpoint Conventions

The supplemental dry eye questionnaire will be collected as shown in Table 6-26.

Table 6-26 Supplemental Dry Eye Questionnaire

| Dry Eye Symptoms Questionnaire | Score |
|---|---|
| In the last 7 days, have you experienced the following symptoms in your right (or | Frequency: |
| left) eye? | • 0=All of the time |
| 1. Dryness | • 1=Most of the time |
| 2. Sensitivity to light | • 2=Half of the time |
| 3. Pain | • 3=Some of the time |
| 4. Decreased or blurred vision | • 4=None of the time |
| 5. Tearing | |
| 6. Experienced feeling like something doesn't belong in your eye | Severity: |
| 7. Secretion or discharge | • 0=Very mild |
| 8. Burning or stinging | • 1=Mild |
| 9. Redness | • 2=Moderate |
| 10. Swelling in the upper eyelid | • 3=Severe |
| 11. Swelling in the lower eyelid | |
| 12. Irritation | • 4=Very severe |
| 13. Grittiness or feeling as if small specks of sand are in your eye | |
| 14. Discomfort | |
| Treatment Satisfaction Questionnaire | |

| Dry Eye Symptoms Questionnaire | Score |
|---|---|
| Taking your entire treatment experience into consideration, if given the choice | 0=Very unlikely |
| again, how likely would you be to repeat the procedure you received in your right | • 1=Unlikely |
| (or left) eye? | • 2=Neither likely or |
| | unlikely |
| | • 3=Likely |
| | • 4=Very likely Mild |

# **6.7 Imputed Value Listing Conventions**

In general, listings will present the actual partial or missing values rather than the imputed values.

# **ALLERGAN**

